CLINICAL TRIAL: NCT02277535
Title: An Email Intervention to Prevent Iatrogenic Malnutrition in the ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daniel Dante Yeh, Trauma and Critical Care Surgeon, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2014P001702
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Malnutrition
Keywords: Malnutrition in the ICU (caloric deficit >4000 kcal or 150 g protein deficit) or >48hrs of admission without receiving nutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- E-mail intervention (Experimental): ICU clinicians caring for patients who have not yet been initiated on nutrition 48 hours after ICU admission will receive a reminder email.
  ICU clinicians caring for patients who accumulate a caloric deficit greater than 4000 calories or 150 g protein deficit will receive a feedback email
  Interventions: Other: Feedback/Reminder email.
- No E-mail intervention (No Intervention): Nutrition status of patients will be assessed but no reminder or feedback emails will be sent

INTERVENTIONS:
Other: Feedback/Reminder email.
  Arms: E-mail intervention

SUMMARY:
This is a quality improvement research project evaluating if a targeted feedback email to clinicians impacts their nutrition delivery in the ICU.

DETAILED DESCRIPTION:
This prospective study looks to determine if a targeted email to clinicians taking care of critically ill patients will allow reduce malnutrition in the Intensive Care Units (ICU). Four ICUs will be included: medical ICU (MICU), coronary care unit (CCU) and two surgical ICUs. The investigators will rotate a 2 month period intervention amongst the aforementioned participating ICUs and follow simultaneous cohorts to evaluate the effect of our intervention (email feedback to treating clinicians) on nutrition delivery in the ICU. After the completion of the intervention, there will be a six-month follow-up of nutritional adequacy to assess the durability of changes in behavior.

ELIGIBILITY:
Inclusion Criteria:

* Clinicians taking care of patients admitted to the ICU within the past 48hrs
* Clinicians taking care of patients in whom enteral nutrition is prescribed

Exclusion Criteria:

* Clinicians taking care of patients in whom enteral nutrition is not prescribed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2014-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Patients started on nutrition within 72 h of ICU admission | After completing the intervention for each ICU (2 months)
  The ICU admission date and EN initiation date will be collected in a data base which will later be analyzed to assess the percentange of patients initiated on EN within 72 hours of admission to the ICU. This will be reported as rates and will be compared amongst intervention and no-intervention arms using Fisher's Exact test or Chi-sq Test